CLINICAL TRIAL: NCT03311399
Title: Using mHealth Technology to Identify and Refer Surgical Site Infections in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Partners in Health (Other)
Responsible Party: Principal Investigator, Robert Riviello, Associate Surgeon, Division of Trauma, Burns and Surgical Critical Care, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016P001943
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Surgical Site Infection
Keywords: Surgical Site Infection; mHealth; Cesarean Section
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Visit (Experimental): Individuals in Arm 1 will be visited at home by the sCHW who will administer the optimized SSI protocol via the mHealth device. Intervention: "SSI Screening Tool used in home visits by CHWs"
  Interventions: Other: SSI Screening Tool used in home visits by CHWs
- Phone Call (Experimental): Individuals in Arm 2 will be phoned by the sCHW who will administer the SSI protocol over the phone. Intervention: "SSI Screening Tool used via phone call follow-up"
  Interventions: Other: SSI Screening Tool used via phone call follow-up
- Standard of Care (No Intervention): Individuals in Arm 3 will not have any additional contact beyond standard of care.

INTERVENTIONS:
Other: SSI Screening Tool used in home visits by CHWs — Individuals in Arm 1 will be visited at home by the sCHW who will administer the optimized SSI protocol via the mHealth device. Following the screening, the sCHWs will use the cell phone to photograph the surgical wound and record the GPS location of the visit.
  Arms: Home Visit
Other: SSI Screening Tool used via phone call follow-up — Individuals in Arm 2 will be phoned by the sCHW who will administer the SSI protocol over the phone.
  Arms: Phone Call

SUMMARY:
The present study aims to examine whether or not the use of mobile Health (mHealth) by community health workers (CHWs) can improve the identification of surgical site infection (SSI) and a timely return to care among patients who undergo cesarean-section surgery at a rural hospital in Rwanda.

DETAILED DESCRIPTION:
Surgical site infections (SSI) are a significant cause of morbidity and mortality worldwide, and particularly in low- and middle-income countries, where geographic and infrastructural barriers often delay or prevent post-operative patients from returning to care. In these settings, rates of SSI can reach 30%. In Rwanda, the current standard of care does not include follow-up of post-operative surgical patients. There, a network of community health workers (CHWs) is employed to provide care and follow-up for pregnant and post-partum women as well as children under five years of age. However, the limited education and existing work load of these workers preclude them from supporting the follow-up of other specialized conditions, such as post-operative patients.

The interventions evaluated in this proposed research seeks to address these gaps. The main aim is to evaluate the impact of the SSI screening protocol, delivered by sCHWs equipped with mHealth support, on the rate of return to care for patients with SSI 10 days post-operation. Two CHW-mHealth interventions will be evaluated. In the first, a sCHW will visit post-operative study participants in their homes to administer the screening protocol prompted by the mobile phone. In the second, a sCHW will call the patient and administer the same screening protocol over the phone. In this phase of the research, 364 patients will be assigned to each of these delivery arms, and the rates of appropriate return to care will be compared to that of 364 patients in a control arm receiving the standard of care (i.e. no additional follow-up). Process indicators also will be reported to describe the feasibility of CHW-mHealth interventions.

Investigators believe that the SSI screening protocol administered via CHW-mHealth interventions can support accurate diagnosis of SSI and refer patients back to the hospital for appropriate follow-up care. The research team's close collaboration with colleagues at the Rwanda Ministry of Health will facilitate the scale-up of the intervention, should it prove efficacious. Results of this study will also inform the development of similar mHealth interventions across other disease areas, allowing CHWs to expand services to other specialized patients in rural African settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients that have undergone cesarean-section surgery at Kirehe District Hospital

Exclusion Criteria:

* Patients from Mahama Refugee Camp will not be asked to participate in follow-up activities due to travel autonomy issues
* Patients that are not residents of Kirehe District
* Patients that have surgery other than cesarean delivery
* Patients that have not been discharged by 7 post-operative days (POD)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with SSI returning to care | by 20 days post-surgery
  The number of patients in each study arm who return to care with a surgical site infection.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Hedt-Gauthier, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Kirehe District Hospital, Kirehe District, Kirehe District, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allegranzi B, Bagheri Nejad S, Combescure C, Graafmans W, Attar H, Donaldson L, Pittet D. Burden of endemic health-care-associated infection in developing countries: systematic review and meta-analysis. Lancet. 2011 Jan 15;377(9761):228-41. doi: 10.1016/S0140-6736(10)61458-4. Epub 2010 Dec 9. PMID 21146207
- [Background] Bagheri Nejad S, Allegranzi B, Syed SB, Ellis B, Pittet D. Health-care-associated infection in Africa: a systematic review. Bull World Health Organ. 2011 Oct 1;89(10):757-65. doi: 10.2471/BLT.11.088179. Epub 2011 Jul 20. PMID 22084514
- [Background] Grimes CE, Bowman KG, Dodgion CM, Lavy CB. Systematic review of barriers to surgical care in low-income and middle-income countries. World J Surg. 2011 May;35(5):941-50. doi: 10.1007/s00268-011-1010-1. PMID 21360305
- [Background] Hsia RY, Mbembati NA, Macfarlane S, Kruk ME. Access to emergency and surgical care in sub-Saharan Africa: the infrastructure gap. Health Policy Plan. 2012 May;27(3):234-44. doi: 10.1093/heapol/czr023. Epub 2011 Mar 26. PMID 21441566
- [Background] Bercion R, Gaudeuille A, Mapouka PA, Behounde T, Guetahoun Y. [Surgical site infection survey in the orthopaedic surgery department of the "Hopital communautaire de Bangui," Central African Republic]. Bull Soc Pathol Exot. 2007 Aug;100(3):197-200. French. PMID 17824315
- [Background] Gottrup F, Melling A, Hollander DA. An overview of surgical site infections: aetiology, incidence and risk factors. EWMA Journal. 2005.
- [Background] Lehman U, Sanders D. Community Health Workers: What do we know about them? The State of the Evidence on Programmes, Activities, Costs and Impact on Health Outcomes Using Community Health Workers. Geneva: World Health Organization, 2007.
- [Background] Mugeni C, Levine AC, Munyaneza RM, Mulindahabi E, Cockrell HC, Glavis-Bloom J, Nutt CT, Wagner CM, Gaju E, Rukundo A, Habimana JP, Karema C, Ngabo F, Binagwaho A. Nationwide implementation of integrated community case management of childhood illness in Rwanda. Glob Health Sci Pract. 2014 Aug 5;2(3):328-41. doi: 10.9745/GHSP-D-14-00080. eCollection 2014 Aug. PMID 25276592
- [Background] Rwanda Health Sector Strategic Plan 2012-2018. Government of Rwanda Ministry of Health. Available online at http://www.moh.gov.rw/fileadmin/templates/Docs/HSSP_III_FINAL_VERSION.pdf.
- [Background] Farmer PE, Nutt CT, Wagner CM, Sekabaraga C, Nuthulaganti T, Weigel JL, Farmer DB, Habinshuti A, Mugeni SD, Karasi JC, Drobac PC. Reduced premature mortality in Rwanda: lessons from success. BMJ. 2013 Jan 18;346:f65. doi: 10.1136/bmj.f65. PMID 23335479
- [Background] Rich ML, Miller AC, Niyigena P, Franke MF, Niyonzima JB, Socci A, Drobac PC, Hakizamungu M, Mayfield A, Ruhayisha R, Epino H, Stulac S, Cancedda C, Karamaga A, Niyonzima S, Yarbrough C, Fleming J, Amoroso C, Mukherjee J, Murray M, Farmer P, Binagwaho A. Excellent clinical outcomes and high retention in care among adults in a community-based HIV treatment program in rural Rwanda. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):e35-42. doi: 10.1097/QAI.0b013e31824476c4. PMID 22156912
- [Background] Franke MF, Kaigamba F, Socci AR, Hakizamungu M, Patel A, Bagiruwigize E, Niyigena P, Walker KD, Epino H, Binagwaho A, Mukherjee J, Farmer PE, Rich ML. Improved retention associated with community-based accompaniment for antiretroviral therapy delivery in rural Rwanda. Clin Infect Dis. 2013 May;56(9):1319-26. doi: 10.1093/cid/cis1193. Epub 2012 Dec 18. PMID 23249611
- [Background] Condo J, Mugeni C, Naughton B, Hall K, Tuazon MA, Omwega A, Nwaigwe F, Drobac P, Hyder Z, Ngabo F, Binagwaho A. Rwanda's evolving community health worker system: a qualitative assessment of client and provider perspectives. Hum Resour Health. 2014 Dec 13;12:71. doi: 10.1186/1478-4491-12-71. PMID 25495237
- [Background] Palazuelos D, Ellis K, Im DD, Peckarsky M, Schwarz D, Farmer DB, Dhillon R, Johnson A, Orihuela C, Hackett J, Bazile J, Berman L, Ballard M, Panjabi R, Ternier R, Slavin S, Lee S, Selinsky S, Mitnick CD. 5-SPICE: the application of an original framework for community health worker program design, quality improvement and research agenda setting. Glob Health Action. 2013 Apr 3;6:19658. doi: 10.3402/gha.v6i0.19658. PMID 23561023
- [Background] Statistical Yearbook. Kigali: National Institute of Statistics of Rwanda, 2014.
- [Background] Mitchell M, Hedt-Gauthier BL, Msellemu D, Nkaka M, Lesh N. Using electronic technology to improve clinical care - results from a before-after cluster trial to evaluate assessment and classification of sick children according to Integrated Management of Childhood Illness (IMCI) protocol in Tanzania. BMC Med Inform Decis Mak. 2013 Aug 27;13:95. doi: 10.1186/1472-6947-13-95. PMID 23981292
- [Background] Mitchell M, Getchell M, Nkaka M, Msellemu D, Van Esch J, Hedt-Gauthier B. Perceived improvement in integrated management of childhood illness implementation through use of mobile technology: qualitative evidence from a pilot study in Tanzania. J Health Commun. 2012;17 Suppl 1:118-27. doi: 10.1080/10810730.2011.649105. PMID 22548605
- [Background] Derenzi B, Borriello G, Jackson J, Kumar VS, Parikh TS, Virk P, Lesh N. Mobile phone tools for field-based health care workers in low-income countries. Mt Sinai J Med. 2011 May-Jun;78(3):406-18. doi: 10.1002/msj.20256. PMID 21598267
- [Background] Mitsunaga T, Hedt-Gauthier B, Ngizwenayo E, Farmer DB, Karamaga A, Drobac P, Basinga P, Hirschhorn L, Ngabo F, Mugeni C. Utilizing community health worker data for program management and evaluation: systems for data quality assessments and baseline results from Rwanda. Soc Sci Med. 2013 May;85:87-92. doi: 10.1016/j.socscimed.2013.02.033. Epub 2013 Mar 1. PMID 23540371
- [Background] Matousek A, Paik K, Winkler E, Denike J, Addington SR, Exe C, Louis RR, Riviello R. Community health workers and smartphones for the detection of surgical site infections in rural Haiti: a pilot study. Lancet. 2015 Apr 27;385 Suppl 2:S47. doi: 10.1016/S0140-6736(15)60842-X. Epub 2015 Apr 26. PMID 26313096
- [Background] Taye M. Wound infection in Tikur Anbessa hospital, surgical department. Ethiop Med J. 2005 Jul;43(3):167-74. PMID 16370548
- [Background] Barie PS, Eachempati SR. Surgical site infections. Surg Clin North Am. 2005 Dec;85(6):1115-35, viii-ix. doi: 10.1016/j.suc.2005.09.006. PMID 16326197
- [Background] Zandbergen PA. Ensuring Confidentiality of Geocoded Health Data: Assessing Geographic Masking Strategies for Individual-Level Data. Adv Med. 2014;2014:567049. doi: 10.1155/2014/567049. Epub 2014 Apr 29. PMID 26556417
- [Derived] Kateera F, Riviello R, Goodman A, Nkurunziza T, Cherian T, Bikorimana L, Nkurunziza J, Nahimana E, Habiyakare C, Ntakiyiruta G, Matousek A, Gaju E, Gruendl M, Powell B, Sonderman K, Koch R, Hedt-Gauthier B. The Effect and Feasibility of mHealth-Supported Surgical Site Infection Diagnosis by Community Health Workers After Cesarean Section in Rural Rwanda: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Jun 8;10(6):e35155. doi: 10.2196/35155. PMID 35675108
- [Derived] Sonderman KA, Nkurunziza T, Kateera F, Gruendl M, Koch R, Gaju E, Habiyakare C, Matousek A, Nahimana E, Ntakiyiruta G, Riviello R, Hedt-Gauthier BL. Using mobile health technology and community health workers to identify and refer caesarean-related surgical site infections in rural Rwanda: a randomised controlled trial protocol. BMJ Open. 2018 May 8;8(5):e022214. doi: 10.1136/bmjopen-2018-022214. PMID 29739786

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03311399/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03311399/ICF_001.pdf